CLINICAL TRIAL: NCT00777920
Title: ABS-LT: A Phase 3, Long-Term, Open Label, Multicenter Safety Study of Ambrisentan in Subjects With Pulmonary Hypertension
Brief Title: Study of Ambrisentan in Participants With Pulmonary Hypertension
Acronym: ABS-LT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-300-0124
Record Dates: First submitted 2008-07-01; First posted 2008-10-22 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ambrisentan (Experimental): Participants will receive ambrisentan 2.5 mg, 5 mg or 10 mg tablet orally once daily until such time as the investigator or participant chooses to stop ambrisentan treatment, ambrisentan becomes commercially available, or the sponsor stops the study.
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Tablet administered orally once daily
  Other Names: Letairis®; Volibris

SUMMARY:
The primary objective of this study is to monitor the long-term safety of ambrisentan in adult participants with pulmonary hypertension. The available ambrisentan doses for this study are 2.5, 5, or 10 mg administered orally once daily. Investigators will be able to adjust ambrisentan dose as clinically indicated. A minimum of 4 weeks between dose adjustments is required. Participants receiving other therapies for pulmonary hypertension that are not contraindicated for concomitant use with ambrisentan are permitted to enroll in this study and continue to receive such therapies. Participants enrolled in this study will receive treatment with ambrisentan until such time as the investigator or participant chooses to stop ambrisentan treatment, ambrisentan becomes commercially available, or the sponsor stops the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women with pulmonary hypertension who are discontinuing a clinical study of ambrisentan due to study closure by the sponsor. Eligible participants are those participating in countries where ambrisentan is not yet commercially available. Participants participating in countries where ambrisentan is commercially available may be eligible if they do not qualify for treatment per the current prescribing information of that country.

Key Exclusion Criteria:

* Participants who have discontinued an ambrisentan clinical study for any other reason than sponsor-initiated study closure are not eligible.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (46):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Atlanta Institute for Medical Research, Inc., Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - BACH Cardiology/Children's Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mary Parkes Asthma Center University of Rochester, Rochester, New York
  - University of Pittsburgh Medical Center Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Lexington Pulmonary and Critical Care Medicine, Lexington, South Carolina
- Argentina (10):
  - Clinica Independencia Munro, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Buenos Aires
  - Sanatorio Otamendi y Miroli, Buenos Aires
  - Hospital Británico de Buenos Aires, Buenos Aires
  - UAI Hospital Universitario, Buenos Aires
  - Instituto de Cardiologia J.F. Cabral, Corrientes
  - Fundación Rusculleda, Córdoba
  - Instituto de Cardiologia Hospital Italiano de Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
  - Hospital Italiano, Rosario
- Australia (2):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Royal Perth Hospital, Perth, Western Australia
- Brazil (6):
  - Instituto de Pneumologia e Pediatria Clínica e Pesquisas LTDA ME, Belo Horizonte
  - UBEA, Hospital Sao Lucas de Pontifícia, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - Universidade do Estado de Sao Paulo - UNIFESP, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo
- Peter Lougheed Centre, Calgary, Alberta, Canada
- Chile (3):
  - Centro de Estudios Cardiologicos Santiago Oriente, Santiago
  - Instituto Nacional del Torax, Santiago
  - Hospital Clinico de la Pontificia Universidad Catolica de Chile, Santiago
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Unidad de Investigacion Clinica en Medicina S.C., Monterrey
- Russia (4):
  - State Medico Stomatologic University, Moscow
  - Russian Cardiology Research Complex, Moscow
  - Almazov's Federal Heart, Blood & Endocrinology Center, Saint Petersburg
  - Pavlov's State Medical University of St. Petersburg, Saint Petersburg
- Ukraine (2):
  - Department of Acute Myocardial Infarction, Kharkiv
  - Department of Propedeutics of Internal Medicine No 1, Kiev

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Argentina, Australia, Brazil, Canada, Chile, Mexico, Russia, Ukraine, and United States. The first participant was screened on 17 November 2008. The last study observation occurred on 11 September 2019.
Pre-assignment Details: 140 participants were screened.
Groups:
- Ambrisentan: Participants received ambrisentan 2.5 mg, 5 mg or 10 mg tablet orally once daily until such time as the investigator or participant chose to stop ambrisentan treatment, ambrisentan became commercially available, or the sponsor stopped the study.
Period: Overall Study
Arm/Group | Ambrisentan
Started | 140
Completed | 90
Not Completed | 50
Not completed — Adverse Event | 39
Not completed — Withdrawal of Consent | 4
Not completed — Lost to Follow-up | 1
Not completed — Investigator's discretion | 1
Not completed — Clinical status did not improve | 1
Not completed — Other, not specified | 4

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were enrolled into the study and received at least one dose of study drug.
Arm/Group | Ambrisentan
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 4
  Race: Black or African American | 5
  Race: White | 126
  Race: Other | 4
Region of Enrollment [Number; unit: participants]
  Argentina | 18
  Australia | 31
  Brazil | 19
  Canada | 2
  Chile | 13
  Mexico | 12
  Russia | 14
  Ukraine | 2
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Associated With Long-Term Exposure to Ambrisentan
Time Frame: First dose date of study drug up to the date of last dose plus 30 days (Maximum: approximately 550 weeks)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 140
percentage of participants | 90.7

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose of study drug up to the date of last dose plus 30 days (Maximum: approximately 550 weeks); All-Cause Mortality: First dose date up to approximately 564 weeks
Description: The Safety Analysis Set included participants who were enrolled into the study and received at least one dose of study drug.
Arm/Group | Ambrisentan
All-Cause Mortality (participants affected / at risk) | 39/140
Serious Adverse Events (participants affected / at risk) | 80/140
Other Adverse Events (participants affected / at risk) | 112/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=140)
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Atrial flutter (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 5
Cardiogenic shock (Cardiac disorders) | 2
Cardiopulmonary failure (Cardiac disorders) | 2
Cor pulmonale (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 13
Deafness unilateral (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 3
Strangulated hernia (General disorders) | 1
Sudden death (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Breast cellulitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Infected fistula (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Pertussis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 12
Respiratory tract infection (Infections and infestations) | 2
Salmonellosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Streptococcal sepsis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vascular device infection (Infections and infestations) | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Burns first degree (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
International normalised ratio increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Device dislocation (Product Issues) | 1
Device malfunction (Product Issues) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Urinary bladder polyp (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 12
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 2
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=140)
Anaemia (Blood and lymphatic system disorders) | 12
Iron deficiency anaemia (Blood and lymphatic system disorders) | 11
Atrial fibrillation (Cardiac disorders) | 9
Palpitations (Cardiac disorders) | 19
Right ventricular failure (Cardiac disorders) | 7
Hypothyroidism (Endocrine disorders) | 8
Cataract (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 9
Chest pain (General disorders) | 9
Fatigue (General disorders) | 16
Oedema peripheral (General disorders) | 41
Bronchitis (Infections and infestations) | 7
Cellulitis (Infections and infestations) | 7
Lower respiratory tract infection (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 10
Pneumonia (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 32
Urinary tract infection (Infections and infestations) | 12
Blood creatinine increased (Investigations) | 7
Gamma-glutamyltransferase increased (Investigations) | 10
Heart sounds abnormal (Investigations) | 10
International normalised ratio increased (Investigations) | 7
Gout (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 19
Headache (Nervous system disorders) | 25
Syncope (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 12
Depression (Psychiatric disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2013-06-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT00777920/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT00777920/SAP_001.pdf